CLINICAL TRIAL: NCT02504710
Title: Kinematic Real-Time Feedback, Obtained by Inertial Sensors, Used to Learn Manual Therapy on Peripherical Joints
Brief Title: Kinematic Real Time Feedback Used to Learn Manual Therapy on Peripherical Joints
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaga (Other)
Responsible Party: Principal Investigator, Dr. Antonio I Cuesta-Vargas, Professor - PhD, University of Malaga
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSF_ISLPerip_Man
Record Dates: First submitted 2015-07-12; First posted 2015-07-22 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2015-07

CONDITIONS: Musculoskeletal Diseases; Complication of Manipulation Procedure; Defective; Learning (Specific)
Keywords: Musculoskeletal Manipulations; Learning; Feedback; Kinematics; Inertial Sensor
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Traditional Learning System (Active Comparator): Traditional systems of manual therapy teaching
  Interventions: Other: Traditional systems of manual therapy teaching
- Kinematic Real-Time Feedback (Experimental): Kinematic real time feedback to learn Manual therapy
  Interventions: Device: Kinematic Real Time Feedback

INTERVENTIONS:
Device: Kinematic Real Time Feedback
  Arms: Kinematic Real-Time Feedback
Other: Traditional systems of manual therapy teaching
  Arms: Traditional Learning System

SUMMARY:
This study will try to analyze the effect of the real-time kinematic feedback (KRTF) to learn manual therapy on peripherical joints comparing the results with the traditional teaching method.

ELIGIBILITY:
Inclusion Criteria:

* undergraduate students with no experience in manual therapy

Exclusion Criteria:

* To have some experience in manual therapy

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-02; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Manipulation time Score | Baseline
  Manipulation time Score: Seconds
Manipulation time Score | One Lesson
  Manipulation time Score: Seconds
Manipulation time Score | One week
  Manipulation time Score: Seconds
Manipulation time Score | Four weeks
  Manipulation time Score: Seconds
Manipulation time Score | Three months
  Manipulation time Score: Seconds
Manipulation time Score | Six Months
  Manipulation time Score: Seconds
Manipulation Displacement Score | Baseline
  Joint Displacement Score: Degrees and centimeter
Manipulation Displacement Score | One Lesson
  Joint Displacement Score: Degrees and centimeter
Manipulation Displacement Score | One week
  Joint Displacement Score: Degrees and centimeter
Manipulation Displacement Score | Four weeks
  Joint Displacement Score: Degrees and centimeter
Manipulation Displacement Score | Three months
  Joint Displacement Score: Degrees and centimeter
Manipulation Displacement Score | Six Months.
  Joint Displacement Score: Degrees and centimeter
Manipulation Mean Velocity Score | Baseline
  Mean Velocity Score: Degrees / seconds and centimeters / seconds
Manipulation Mean Velocity Score | One Lesson
  Mean Velocity Score: Degrees / seconds and centimeters / seconds
Manipulation Mean Velocity Score | One week
  Mean Velocity Score: Degrees / seconds and centimeters / seconds
Manipulation Mean Velocity Score | Four weeks
  Mean Velocity Score: Degrees / seconds and centimeters / seconds
Manipulation Mean Velocity Score | Three months
  Mean Velocity Score: Degrees / seconds and centimeters / seconds
Manipulation Mean Velocity Score | Six months.
  Mean Velocity Score: Degrees / seconds and centimeters / seconds
Manipulation Maximal Velocity Score | Baseline
  Maximal Velocity Score: Degrees / seconds and centimeters / seconds
Manipulation Maximal Velocity Score | One Lesson
  Maximal Velocity Score: Degrees / seconds and centimeters / seconds
Manipulation Maximal Velocity Score | One week
  Maximal Velocity Score: Degrees / seconds and centimeters / seconds
Manipulation Maximal Velocity Score | Four weeks
  Maximal Velocity Score: Degrees / seconds and centimeters / seconds
Manipulation Maximal Velocity Score | Three months
  Maximal Velocity Score: Degrees / seconds and centimeters / seconds
Manipulation Maximal Velocity Score | Six months.
  Maximal Velocity Score: Degrees / seconds and centimeters / seconds
Manipulation Mean Acceleration Score | Baseline
  Mean Acceleration Score: (Degrees / seconds)2 and (centimeters / seconds)2
Manipulation Mean Acceleration Score | One Lesson
  Mean Acceleration Score: (Degrees / seconds)2 and (centimeters / seconds)2
Manipulation Mean Acceleration Score | One week
  Mean Acceleration Score: (Degrees / seconds)2 and (centimeters / seconds)2
Manipulation Mean Acceleration Score | Four weeks
  Mean Acceleration Score: (Degrees / seconds)2 and (centimeters / seconds)2
Manipulation Mean Acceleration Score | Three months
  Mean Acceleration Score: (Degrees / seconds)2 and (centimeters / seconds)2
Manipulation Mean Acceleration Score | Six months.
  Mean Acceleration Score: (Degrees / seconds)2 and (centimeters / seconds)2
Manipulation Maximal Acceleration Score | Baseline
  Maximal acceleration Score: (Degrees / seconds)2 and (centimeters / seconds)2
Manipulation Maximal Acceleration Score | One Lesson
  Maximal acceleration Score: (Degrees / seconds)2 and (centimeters / seconds)2
Manipulation Maximal Acceleration Score | One week
  Maximal acceleration Score: (Degrees / seconds)2 and (centimeters / seconds)2
Manipulation Maximal Acceleration Score | Four weeks
  Maximal acceleration Score: (Degrees / seconds)2 and (centimeters / seconds)2
Manipulation Maximal Acceleration Score | Three months
  Maximal acceleration Score: (Degrees / seconds)2 and (centimeters / seconds)2
Manipulation Maximal Acceleration Score | Six months.
  Maximal acceleration Score: (Degrees / seconds)2 and (centimeters / seconds)2

CONTACTS AND LOCATIONS:
Locations (1):
- Antonio I Cuesta-Vargas, Málaga, Málaga, Spain

REFERENCES:
- [Derived] Trinidad-Fernandez M, Gonzalez-Molina F, Roldan-Jimenez C, Vaes P, Gonzalez-Sanchez M, Cuesta-Vargas AI. New learning technique based on real-time kinematic feedback from an inertial sensor for manual therapy in shoulder joint: a randomised trial. BMC Med Educ. 2024 Sep 11;24(1):992. doi: 10.1186/s12909-024-05649-y. PMID 39261790
- [Derived] Gonzalez-Sanchez M, Ruiz-Munoz M, Avila-Bolivar AB, Cuesta-Vargas AI. Kinematic real-time feedback is more effective than traditional teaching method in learning ankle joint mobilisation: a randomised controlled trial. BMC Med Educ. 2016 Oct 6;16(1):261. doi: 10.1186/s12909-016-0789-8. PMID 27716215